CLINICAL TRIAL: NCT02609542
Title: Coding and Memorisation of Phonologic Information Among Preschool and School Children With Oral Language Developement Disorder.
Brief Title: Memorisation of Phonologic Information Among Children With Oral Language Developement Disorder
Acronym: MEMENTO
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0029
Record Dates: First submitted 2015-08-04; First posted 2015-11-20 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Language Development Disorders
Keywords: oral language; STOL; memory; eye tracking
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- STOL group: STOL children will be recruited in the neuropediatric unit at the GHICL in Lille. Children will be followed and we will determine if capacities of verbal memory of the children presenting STOL diagnosed at an early stage of their development (before 6 years) are predictive of the evolution of the disorder according to their cognitive profile and more specifically, their language profile as well as their tests performances. The participants' eye movements ( visual world paradigm or eye tracking) will be recorded in order to determine the interplay between linguistic and visual information processing.
  Patients with a persistent STOL will be identified at the end of the follow up.
  Interventions: Other: Eye Tracking
- Control group: Children with no language development disorder willing to participate in the study will be recruited at school. The participants' eye movements ( visual world paradigm or eye tracking) will be recorded in order to determine the interplay between linguistic and visual information processing.
  Interventions: Other: Eye Tracking

INTERVENTIONS:
Other: Eye Tracking — Eye tracker will allows the recording of various information concerning eye fixation (number, duration, location) and saccadic eye movement (speed, range, number, duration) in order to determine the interplay between linguistic and visual information processing during tests performance
  Other Names: visual world paradigm

SUMMARY:
The disorder of oral language development is defined by the delay in language acquisition in children who possess efficient auditory acuity and normal non verbal intellect.

The diversity of language developement disorders depends either in the expressive level or in the receptive level leading to divers syndromes and symptoms. These syndromes and symptoms are regrouped under the name of STOL (Specific Troubles of Oral Language).

In the current project the visual exploitation and learning capability of children presenting a STOL condition will be compared to patients with a normal development. The investigator's hypothesis is as follows: STOL patients for whom the STOL disorder is reduced between 4 and 7 years of age will present a better performance at verbal memorisation, compared to patients with a persistent STOL condition after the age of 6.

ELIGIBILITY:
Inclusion Criteria for STOL patients:

* Child aged between 45 and 95 months at inclusion
* A score > or equal to 5 percentile on the non verbal intelligence test (PM47)
* Patient diagnosed with STOL by the neuropediatric medical team
* Coverage of the social insurance
* Consent form signed by the parents or the legal representative of the child
* Normal or corrected sight
* Normal hearing

Inclusion Criteria for control patients:

* Child aged between 45 and 95 months on the day of inclusion
* A score > or equal to 5 percentile on the non verbal intelligence test (PM47)
* Child who did not receive any speech therapy
* Coverage of the social insurance
* Consent form signed by the parents or the legal representative of the child
* Normal or corrected sight
* Normal hearing

Exclusion Criteria for STOL patients:

* Mother language other than French
* Score < to 5 percentile on the non verbal intelligence test (PM47)
* Child with pervasive developmental disorder

Exclusion Criteria for control patients:

* Mother language other than French
* Score < to 5 percentile on the non verbal intelligence test (PM47)
* Child who received speech therapy

Ages: 45 Months to 95 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: STOL children between 45 and 95 months of age at inclusion recruited at the neuropediatric consultation and control children of the same age recruited at schools
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2014-03; Primary Completion 2023-05 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in the score associated to speech-language outcome measured by a scale grouping results of different questionnaires | 0,12, 24 months
  We will determine if capacities of verbal memory of the children presenting STOL diagnosed at an early stage of their development (before 6 years) are predictive of the evolution of the disorder according to their cognitive profile and more specifically, their language profile as well as their tests performances. To measure the speech language outcome is necessary to take in consideration the score of more than one test performance.

SECONDARY OUTCOMES:
Changes from baseline in the Raven's Progressive Matrices (RPM) test | 0,12, 24 months
  Raven's Progressive Matrices (RPM) is a test often used in educational settings that is comprised of 60 multiple choice questions. This is a nonverbal test in that the questions are comprised of visual patterns. RPM measures the ability to think clearly about complex ideas and the ability to store and recall information.
Changes from baseline in the Peabody Picture Vocabulary Test | 0,12, 24 months
  The Peabody Picture Vocabulary Test measures an individual's receptive (hearing) vocabulary and provides, at the same time, a quick estimate of verbal ability or scholastic aptitude.
Changes from baseline in the number repetition test | 0,12, 24 months
Changes from baseline in the sentences repetition test | 0,12, 24 months
Changes from baseline in the non-words repetition test | 0,12, 24 months
Changes from baseline in the children's eye tracking | 0,12, 24 months
  It is done in order to determine if their is a relation between the evolution of processes involved in verbal memorisation (cognitive mechanisms in charge of data processing).
  Eye tracker will allow the recording of information regarding eye fixation (number, duration, location) and saccadic eye movements (speed, range, number, duration) in order to determine the interplay between linguistic and visual information processing during test performances.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Fleurion, Psychologist, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille
Locations (1):
- Hôpital St Vincent-de-Paul (GHICL), Lille, Hauts-de-France, France